CLINICAL TRIAL: NCT02040129
Title: Reduction of Corneal Astigmatism With Toric Intraocular Lens Implantation : Early Results in Patients With Congenital Cataract
Brief Title: Reduction of Corneal Astigmatism With Toric Intraocular Lens Implantation in Congenital Cataract
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kyungpook National University Hospital (Other)
Responsible Party: Principal Investigator, Bo Young Chun, Department of Ophthalmology, School of medicine, Kyungpook National University, Kyungpook National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KNUH2014-01
Record Dates: First submitted 2014-01-16; First posted 2014-01-20 (Estimated); Last update posted 2014-01-20 (Estimated); Status verified 2014-01

CONDITIONS: Congenital Cataract

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Acrysof toric IOL (Experimental): Acrysof Toric intraocular lens in congenital cataract
  Interventions: Device: Acrysof Toric IOL

INTERVENTIONS:
Device: Acrysof Toric IOL — Lens implantation following cataract surgery

SUMMARY:
This study was conducted to evaluate changes of reduction of corneal astigmatism with toric intraocular lens(IOL) in congenital cataract.

DETAILED DESCRIPTION:
This retrospective study included 6 eyes from 4 patients (mean age 7.2 years) with congenital cataract who had an astigmatism of 2.5 to 4.0 D prior to cataract surgery. Review of preoperative and postoperative visual acuity (UCVA), refraction, toric axis was performed.

ELIGIBILITY:
Inclusion Criteria:

* Children less than 14 years
* Congenital cataract at initial visit
* Symmetrical keratometric astigmatism more than 2.0 D

Exclusion Criteria:

* Microcornea (horizontal corneal diameter less than 9.5mm-asper that particular age)
* Corneal pathology
* Keratoconus
* Irregular astigmatism

Ages: 1 Year to 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 4 (Actual)
Dates: Start 2009-01; Primary Completion 2009-01 (Actual); Study Completion 2009-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline in astigmatism after cataract surgery at 24 months | preop, 3,6,12,24 month postop
  Measurement of refraction after cataract surgery was performed.

SECONDARY OUTCOMES:
Change from baseline in quality of vision after cataract surgery at 24 months. | preop, 3,6,12,24 months postop
  Measurement of visual acuity after cataract surgery was performed.

CONTACTS AND LOCATIONS:
Overall Officials: Bo Young Chun, M.D, Principal Investigator — Kyungpook National University Hospital
Locations (1):
- Bo Young Chun, M.D., Daegu, Kyungsangpookdo, South Korea